CLINICAL TRIAL: NCT00351351
Title: Randomized Control Trial Comparing Dual Probe Ultrasonic Lithotripsy to a Single Probe Ultrasonic Lithotripsy
Brief Title: Trial Comparing Dual Probe Ultrasonic Lithotripsy to a Single Probe Ultrasonic Lithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana Kidney Stone Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-035
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Results first posted 2013-02-20 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2013-02

CONDITIONS: Kidney Stones
Keywords: Kidney Stones; Renal Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Cyberwand
  Interventions: Device: Cyberwand
- B (Active Comparator): Currently available lithotripsy technology
  Interventions: Device: single probe ultrasonic

INTERVENTIONS:
Device: Cyberwand — FDA approved - dual probe intracorporeal lithotrite
  Arms: A
Device: single probe ultrasonic — FDA-approved - single probe ultrasonic
  Arms: B

SUMMARY:
Percutaneous nephrolithotomy (PNL), in conjunction with intracorporeal lithotripsy, allows for the rapid removal of any kidney stone regardless of size. Currently, the choice of intracorporeal lithotripters includes ultrasonic, pneumatic, and combined ultrasonic/pneumatic energy sources. Recently, a novel dual probe design as been introduced by Cybersonics of Erie, Pennsylvania. This dual probe intracorporeal lithotrite is called the Cyberwand, and is composed of a fixed inner probe vibrating at an ultrasonic frequency with an outer probe vibrating at about 1,000 Hz. As this new design has the potential to revolutionize intracorporeal lithotripsy, we intend to compare this novel technology to currently available lithotripsy technology in a randomized clinical trial.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PNL) is used to remove large and complex stones from the upper urinary tract. Intracorporeal lithotripsy is an integral part of PNL. Commercially available intracorporeal lithotripsy modalities include ultrasonic, pneumatic, and combined ultrasonic and pneumatic models. Each modality has its inherent advantages and disadvantages. Ultrasonic lithotrites are capable of fragmenting stones while concomitantly suctioning out fragments. Unfortunately some stones are hard enough to resist fragmentation from ultrasonic lithotripsy. Pneumatic lithotrites are able to fragment all stones regardless of hardness, but this modality is unable to suction out stone pieces at the same time fragmentation is occurring. The newest lithotrite which combines both ultrasonic and pneumatic components is capable of fragmenting any stone, but also has some inherent limitations. The handpiece of the lithotripsy device is somewhat cumbersome, the suction component can clog, and the device has overheated at the maximal settings (Kuo et al). Current intracorporeal lithotrites, while functional, can certainly be improved.

Recently, a novel dual probe design has been introduced by Cybersonics of Erie, PA. This dual probe intracorporeal lithotrite is called the Cyberwand and is composed of a fixed inner probe vibrating at an ultrasonic frequency with an outer probe vibrating at about 1,000 Hz. As this new design has the potential to revolutionalize intracorporeal lithotripsy, we intend to compare this novel technology to currently available lithotripsy technology in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient of Methodist Urology in Indianapolis, IN
* Undergoing percutaneous nephrolithotomy for calculi greater than 2 cm
* Age 18 years or older
* Stone easily visible/measurable on kidney, ureters and bladder (KUB) or computed tomography (CT) scan preoperatively

Exclusion Criteria:

* Radiolucent stones
* Size of largest stone less than 2 cm
* Pregnancy
* Inability to give informed consent
* Multiple percutaneous access anticipated
* Active urinary tract infection
* Recent (within last 3 months) extracorporeal shock wave lithotripsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E. Lingeman, MD, Principal Investigator — Methodist Urology
Locations (7):
- United States (5):
  - Northwestern University Dept. of Urology, Chicago, Illinois
  - Methodist Hospital, Indianapolis, Indiana
  - John's Hopkins University, Baltimore, Maryland
  - Duke University, Durham, North Carolina
  - University of Wisconsin, Madison, Wisconsin
- Canada (2):
  - Vancouver Hospital, Vancouver, British Columbia
  - University of Western Ontario - St. Joseph's Hospital, London, Ontario

REFERENCES:
- [Background] Kuo RL, Paterson RF, Siqueira TM Jr, Evan AP, McAteer JA, Williams JC Jr, Lingeman JE. In vitro assessment of lithoclast ultra intracorporeal lithotripter. J Endourol. 2004 Mar;18(2):153-6. doi: 10.1089/089277904322959789. PMID 15072622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing percutaneous nephrolithotomy with a target stone size greater than 2cm
Groups:
- Cyberwand: Cyberwand
  Cyberwand : FDA approved - dual probe intracorporeal lithotrite
- Currently Available Lithotripsy Technology: Currently available lithotripsy technology
  single probe ultrasonic : FDA-approved - single probe ultrasonic
Period: Overall Study
Arm/Group | Cyberwand | Currently Available Lithotripsy Technology
Started | 34 | 36
Completed | 25 | 32
Not Completed | 9 | 4
Not completed — surgical access pbs; device issues | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Currently Available Lithotripsy Techology: Currently available lithotripsy technology
  single probe ultrasonic : FDA-approved - single probe ultrasonic
- Total: Total of all reporting groups
Arm/Group | Cyberwand | Currently Available Lithotripsy Techology | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 31 | 59
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 20 | 22 | 42
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50
  Canada | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Kidney Stone Clearance Rate
Description: stone clearance rate calculated in mm^2/min per protocol specification
Time Frame: 6 months
Population: Sample size calculations were performed using a two-sided Student's t-test with a power of 90% and a significance level of α = 0.05
Measure: Mean (Full Range); unit: mm^2/min
Arm/Group | Cyberwand | Currently Available Lithotripsy Techology
Number analyzed (Participants) | 25 | 32
mm^2/min | 61.9 [6.1 to 222.69] | 75.8 [9.16 to 551.9]

ADVERSE EVENTS:
Arm/Group | Cyberwand | Currently Available Lithotripsy Technology
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 10/34 | 15/36
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyberwand (N=34) | Currently Available Lithotripsy Technology (N=36)
fever (Infections and infestations) | 0 (0) | 3 (3)
hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
perinephric haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
persistent flank pain (General disorders) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
respiratory difficulty (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
discharged home with nephrostomy tube (Renal and urinary disorders) | 4 (4) | 7 (7)

LIMITATIONS AND CAVEATS:
Multiple surgeons were involved,thus subtle differences in PCNL technique existed between sites. Some surgeons may have defined the stone removal time differently.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No